CLINICAL TRIAL: NCT06563024
Title: Prospective Investigation in the Utility of Multiparametric 18F-FET PET/CT in the Management of Glioma: Application of PET Radiomics
Brief Title: 18F-FET PET/CT in the Management of Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB108-262-A
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Glioma
Keywords: Glioma, 18F-FET, PET
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FET PET (Experimental): The study participants receive the 18F-FET PET scan.
  Interventions: Device: 18F-FET PET/CT

INTERVENTIONS:
Device: 18F-FET PET/CT — The enrolled patients receive the 18F-FET PET/CT.

SUMMARY:
O-(2-[18F]-fluoroethyl)-L-tyrosine (FET) is a tracer for positron emission tomography (PET). The Response Assessment in Neuro-Oncology (RANO) working group has officially recommended 18F-FET PET in the management of patients with brain glioma. Recently, the utility of 18F-FET PET in the diagnosis of fresh and residual gliomas has been reported by several investigators. But clinical usefulness of radiomics parameters has not been explored thoroughly in glioma patients. 18F-FET PET has been widely used in clinical studies or routine service in Europe, America, Mainland China, or Japan. However, 18F-FET PET is still not available in Taiwan. In this context, the investigator propose this study to explore the role of multiparametric 18F-FET PET imaging for glioma in Taiwan, with the emphasis in radiomics analysis.

DETAILED DESCRIPTION:
Study background:

O-(2-[18F]-fluoroethyl)-L-tyrosine (FET) is a tracer for positron emission tomography (PET). The Response Assessment in Neuro-Oncology (RANO) working group has officially recommended 18F-FET PET in the management of patients with brain glioma. Recently, the utility of 18F-FET PET in the diagnosis of fresh and residual gliomas has been reported by several investigators. But clinical usefulness of radiomics parameters has not been explored thoroughly in glioma patients. 18F-FET PET has been widely used in clinical studies or routine service in Europe, America, Mainland China, or Japan. However, 18F-FET PET is still not available in Taiwan. In this context, the investigator propose this study to explore the role of multiparametric 18F-FET PET imaging for glioma in Taiwan.

Materials and methods:

1. During the pre-treatment work-up, the study participants undergo an 18F-FET PET/CT scan. In addition, other routine examinations, including MRI with and without contrast enhancement, are performed.
2. After a definitive diagnosis of primary/recurrent glioma is confirmed, subjects begin treatment (surgery, radiation therapy, chemotherapy, etc.). Within 3 to 6 months after completing treatment, the study subjects undergo a second 18F-FET PET/CT scan for response evaluation, along with a follow-up MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary or recurrent brain tumors confirmed by pathological examination or imaging studies.
2. The ability to provide written informed consent and receive the scheduled scan.

Exclusion Criteria:

1. Woman with pregnancy or during lactation.
2. Unsuitable for PET scans, such as those with claustrophobia or inability to lie flat.
3. Unable to sign the informed consent form.
4. Patients with a second primary tumor.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival is measured from the date of diagnosis to the date of death, or censored at last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chieh Chan, Study Director — Hualien Tzu Chi General Hospital
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan SC, Chiu TL, Ng SH, Kao HW, Tsai ST, Liu SH. 18F-FET PET/CT can aid in diagnosing patients with indeterminate MRI findings for brain tumors: a prospective study. Ann Nucl Med. 2025 Apr;39(4):342-352. doi: 10.1007/s12149-024-02005-4. Epub 2024 Nov 26. PMID 39589672